CLINICAL TRIAL: NCT07288892
Title: Effects of Pulsed Electromagnetic Field Therapy on Sport Performance and Recovery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanyang Technological University (Other)
Collaborators: QuantumTX Pte Ltd (Network)
Responsible Party: Principal Investigator, Kong Pui Wah, Associate Professor, Nanyang Technological University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB-2025-575
Record Dates: First submitted 2025-11-16; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Sport Performance; Sport Recovery; Athlete
Keywords: PEMF; Sport; Performance; Recovery; Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active PEMF Group (Experimental): The active PEMF group will receive 8 weeks of active pulsed electromagnetic field therapy.
  Interventions: Device: Active Pulsed Electromagnetic Field Therapy
- Sham PEMF Group (Sham Comparator): The sham PEMF group will receive 8 weeks of sham pulsed electromagnetic field therapy.
  Interventions: Device: Sham Pulsed Electromagnetic Field Therapy

INTERVENTIONS:
Device: Active Pulsed Electromagnetic Field Therapy — The experimental group will receive active Pulsed Electromagnetic Field (PEMF) therapy twice weekly for 8 weeks, for a total of 16 sessions. Participants will sit comfortably in a chair with their legs placed inside the solenoid of the PEMF device. The active PEMF settings are 1.2 milliTesla (mT) at 50 Hertz (Hz). Each PEMF session will last 20 minutes, with 10 minutes of active PEMF exposure per leg.
  Arms: Active PEMF Group
Device: Sham Pulsed Electromagnetic Field Therapy — The control group will receive sham Pulsed Electromagnetic Field (PEMF) therapy twice weekly for 8 weeks, for a total of 16 sessions. Participants will sit comfortably in a chair with their legs placed inside the solenoid of the PEMF device. The sham PEMF settings are 0 milliTesla (mT) at 0 Hertz (Hz). Each PEMF session will last 20 minutes, with 10 minutes of sham PEMF exposure per leg.
  Arms: Sham PEMF Group

SUMMARY:
The goal of this clinical trial is to learn if pulsed electromagnetic field (PEMF) therapy works to improve sports performance and recovery in athletes. The main questions it aims to answer are:

* Does PEMF therapy enhance participants' performance during exercise?
* Does PEMF therapy enhance recovery in participants after exercise? Researchers will compare active PEMF therapy to sham PEMF therapy (using the same device for both, but without any electromagnetic fields) to see if active PEMF therapy is effective in improving sports performance and recovery.

Participants will:

* Receive active pulsed electromagnetic field therapy or sham pulsed electromagnetic field therapy twice a week for 8 weeks.
* Visit the laboratory at baseline, 8 weeks, and 12 weeks for sports performance and recovery assessments.

DETAILED DESCRIPTION:
This is a prospective, randomised, double-blind, placebo-controlled superiority trial with two parallel groups and a 1:1 allocation ratio investigating the effects of PEMF therapy on athletes. Participants will be recruited from the Physical Education and Sports Science Department at the National Institute of Education, Nanyang Technological University in Singapore. Researchers will monitor sports performance and recovery outcomes during baseline assessment and at the 8- and 12-week follow-ups after the start of Pulsed Electromagnetic Field (PEMF) therapy. The PEMF therapy will last for 8 weeks, with the final assessment scheduled at week 12. The outcomes measured at 8 weeks will reflect the short-term effects, while the final time point may indicate the carry-over effects of PEMF therapy on athletes.

The PEMF therapy will be administered using a commercial device (QuantumTX Pte). The delivery of PEMF to the leg will not produce heat or cause any sensation, which allows the participants to be blinded to the treatment. Participants in the control group will receive sham exposure with the same PEMF device. Each leg will undergo either active PEMF therapy or sham PEMF therapy for 10 minutes per session, with the treatment administered twice weekly for 8 weeks, resulting in a total of 16 sessions. The PEMF device will be activated by the Radiofrequency Identification (RFID) card, which will be coded to deliver either the active or sham PEMF treatment. The PEMF therapy procedure will be as follows: The participant will be seated in a 90° position on a chair, and the entire quadriceps muscle will be placed within the solenoids of the PEMF device. When active, the device delivered uniform 1.2 mT, 50 Hz PEMFs to each quadriceps muscle for 10 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Exercise at least twice a week in the past 3 months
* Perform resistance training 1-3 times per week in the past 3 months.
* Have competed in at least two matches / events in the past one year (e.g. heat and final are counted as two events).

Exclusion Criteria:

* History of fracture or surgery over the past year.
* History of musculoskeletal injury in the last 3 months that required more than 7 days of rest.
* Currently experiencing any injury, discomfort and/or pain at the time of study.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Wingate anaerobic test rate of fatigue | From enrollment to the end of treatment at 8 weeks, and a 12-week follow-up
  The Wingate anaerobic test involves a 30-second all-out cycling effort performed while stationary. Participants pedal as fast as possible against a standardised resistance for 30 seconds. The percentage decline in power output is calculated from the peak power to the lowest power during the test. It measures how quickly an individual fatigues during intense anaerobic exercise and their capacity to sustain high power output.
Blood lactate level | From enrollment to the end of treatment at 8 weeks, and a 12-week follow-up
  Finger-prick blood sampling for lactate levels will be performed at 4 time points (baseline and 5, 15, and 30 min after the Wingate anaerobic test).

SECONDARY OUTCOMES:
Wingate anaerobic test peak power | From enrollment to the end of treatment at 8 weeks, and a 12-week follow-up
  The Wingate anaerobic test involves a 30-second all-out cycling effort performed at a stationary position. Participants will pedal as fast as possible against a standardised resistance for 30 seconds. The highest power output achieved during the 30-second Wingate anaerobic test will be recorded as the peak power in Watts.
Wingate anaerobic test mean power | From enrollment to the end of treatment at 8 weeks, and a 12-week follow-up
  The Wingate anaerobic test involves a 30-second all-out cycling effort performed at a stationary position. Participants will pedal as fast as possible against a standardised resistance for 30 seconds. The average power output achieved during the 30-second Wingate anaerobic test will be recorded as the mean power in Watts.
Skeletal muscle mass | From enrollment to the end of treatment at 8 weeks, and a 12-week follow-up
  Skeletal muscle mass in kilograms will be assessed using the InBody Body Composition Analyser while standing. Skeletal muscle mass specifically relates to muscles that can grow through training.
Muscle stiffness | From enrollment to the end of treatment at 8 weeks, and a 12-week follow-up
  Muscle stiffness of the vastus lateralis will be assessed using the MyotonPRO Digital Palpation Device at rest.
Muscle oxygen saturation | From enrollment to the end of treatment at 8 weeks, and a 12-week follow-up
  Muscle oxygen saturation of the vastus lateralis will be measured using Near-Infrared Spectroscopy (NIRS) before, during, and after the Wingate anaerobic test.
Muscle activity | From enrollment to the end of treatment at 8 weeks, and a 12-week follow-up
  Muscle activity of the vastus lateralis will be recorded using surface electromyography (EMG) during the Wingate anaerobic test.
Strength | From enrollment to the end of treatment at 8 weeks, and a 12-week follow-up
  Strength will be measured using the isometric mid-thigh pull test. Participants will pull against a fixed metal chain while standing on the back extension dynamometer platform. The dynamometer will record the maximum force exerted.

CONTACTS AND LOCATIONS:
Overall Officials: Pui Wah KONG, PhD, Principal Investigator — Nanyang Technological University
Locations (1):
- Human Bioenergetics Laboratory, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be shared upon reasonable requests.

REFERENCES:
- See also: Pulsed Electromagnetic Field Therapy — https://www.mitocharge.com/